CLINICAL TRIAL: NCT05940324
Title: Examining Mu Opioid Mechanisms of Ketamine's Rapid Effects in OCD (MKET2)
Acronym: MKET2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 70954; 1R01MH133553-01 (NIH)
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Ketamine; Naltrexone; MRI; Brain Imaging; OCD symptoms; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine; Naltrexone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized with a 1:1 allocation to either IV ketamine + oral placebo or IV ketamine + oral opioid antagonist naltrexone
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ketamine + Naltrexone (Experimental): OCD patients in this arm will receive 0.5mg/kg of ketamine - one single infusion. fMRI will be acquired before, during, and after infusion.
  Oral naltrexone 50 mg will be administered before the infusion.
  Interventions: Drug: Ketamine; Drug: Naltrexone Pill
- Ketamine + Placebo (Placebo Comparator): OCD patients in this arm will receive 0.5mg/kg of ketamine - one single infusion. fMRI will be acquired before, during, and after infusion.
  An oral inactive placebo will be administered before the infusion.
  Interventions: Drug: Ketamine; Other: Placebo pill
- Healthy Volunteers (No Intervention): Healthy volunteers will have one fMRI scan visit.

INTERVENTIONS:
Drug: Ketamine — Ketamine is an FDA-approved dissociative anesthetic.
  Other Names: Ketamine Hydrochloride; Ketalar
  Arms: Ketamine + Naltrexone; Ketamine + Placebo
Drug: Naltrexone Pill — Naltrexone is an oral opioid antagonist approved by the Food and Drug Administration (FDA) to treat both alcohol use disorder (AUD) and opioid use disorder (OUD)
  Other Names: Naltrexone
  Arms: Ketamine + Naltrexone
Other: Placebo pill — An oral inactive placebo pill will be administered to preserve the blinded nature of the study.
  Arms: Ketamine + Placebo

SUMMARY:
The purpose of this study is to understand how ketamine works in the brain to bring about a reduction in OCD symptoms.

DETAILED DESCRIPTION:
The proposed mechanistic trial would be the first to probe the role of ketamine's opioid properties in modulating fronto-striatal circuitry and bringing about reduction of OCD symptoms.

ELIGIBILITY:
Eligibility Criteria for Participants with OCD:

Inclusion Criteria:

* Ages 18-65
* Meet the criteria for OCD diagnosis
* Failed at least 1 prior trial of standard first-line OCD treatment
* Agree to the following lifestyle modifications: comply with requirements for fasting prior to the Experimental Session, not enroll in any other interventional clinical trials during the duration of the study, and commit to medication study procedures.
* Able to provide informed consent

Exclusion Criteria:

* prior naltrexone or ketamine use/exposure
* Any current or past medical/psychiatric condition that makes participation unsafe in the opinion of the investigator or study physician
* Pregnant or nursing, or able to become pregnant and are not practicing an effective means of birth control
* the presence of metal in the body that is contraindicated for MRI scans

Eligibility Criteria for Healthy Volunteers:

Inclusion Criteria:

* Ages 18-65
* Able to provide informed consent

Exclusion Criteria:

* current or past use of psychotropic medication
* pregnant or nursing females
* the presence of metal in the body that is contraindicated for MRI scans

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change in the severity of OCD symptoms as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Baseline (Visit 2) to Post Infusion fMRI scan (Visit 4; Day 1), up to 1 week
  Change in OCD severity is measured by the YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response is defined as at least a 35% reduction on the YBOCS.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry & Behavioral Sciences, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No